CLINICAL TRIAL: NCT05492305
Title: Effect of Glucagon-like Peptide 1 (GLP1) Receptor Agonists on Mental Health in Patients With Obesity and Type 2 Diabetes (T2D): a Mixed Methods Study
Brief Title: Glucagon-like Peptide 1 (GLP1) Receptor Agonists and Mental Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Aureliane Pierret, Principle investigator, King's College London
Other Study IDs: 314639
Record Dates: First submitted 2022-08-03; First posted 2022-08-08 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus; Obesity; Mental Health Issue
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Treatment with any GLP1 receptor agonist e.g. liraglutide, semaglutide, dulaglutide for either obesity or type 2 diabetes mellitus

SUMMARY:
This study is investigating the effect of a medication called glucagon-like peptide 1 (GLP1) receptor agonists on mental health. GLP1 receptor agonists are a type of medication that are used to treat obesity and type 2 diabetes (T2D). Obesity and T2D are very common health conditions, and research has shown that people living with obesity and T2D are more likely to experience mental health disorders. Some recent research has suggested that GLP1 receptor agonists might help with mental health problems such as depression and binge eating disorder, and the investigators want to expand on this in this study. The investigators will be recruiting patients from community diabetes services, and tier 3 weight management services in South East London. Patients will be eligible if they are starting on GLP1 receptor agonists for the management of either T2D or obesity. The study is a mixed methods, longitudinal observations study with two components - a quantitative and a qualitative aspect. Firstly, the investigators will be interviewing patients before and 12-16 weeks after starting the medication, using short questionnaires which asks participants about different mental health symptoms that they may be experiencing. The investigators will use this information to see if there are any objective changes in mental health after taking GLP1 receptor agonists. Secondly, the investigators will be conducting a longer semi-structured interview after the second set of short questionnaires (at 12-16 weeks after starting GLP1 receptor agonist), asking about patient's experiences of taking the medication and how it has affected their mental health and general wellbeing. The investigators will qualitatively analyse this data to determine the subjective effect of GLP1 receptor agonists on mental health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* being commenced on a glucagon-like peptide 1 (GLP1) receptor agonist for management of either for obesity or type 2 diabetes
* least 18 years of age
* able to consent, speak and read in fluent English.

Exclusion Criteria:

* not able to consent, speak and read in fluent English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being commenced on GLP1 receptor agonist for management of either for obesity or type 2 diabetes, according to the NICE guidelines for these indications.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
subjective effect of GLP1 receptor agonist on mental health | 12-16 weeks
  qualitative analysis of the subjective effect of GLP1 receptor agonist on mental health in patients with diabetes and obesity (determined at stage 2 using the semi-structured interview)

SECONDARY OUTCOMES:
subjective effect of GLP1 receptor agonist on general wellbeing | 12-16 weeks
  qualitative analysis of the subjective effect of GLP1 receptor agonist on general wellbeing (determined at stage 2 using the semi-structured interview)
subjective effect of GLP1 receptor agonist on eating behaviours | 12-16 weeks
  qualitative analysis of the subjective effect of GLP1 receptor agonist on eating behaviours (determined at stage 2 using the semi-structured interview)
subjective effect of GLP1 receptor agonist on binge eating, if present | 12-16 weeks
  qualitative analysis of the subjective effect of GLP1 receptor agonist on binge eating, if present (determined at stage 2 using the semi-structured interview)
mean change in patient health questionnaire 9 (PHQ9) score with GLP1 receptor agonist over 12-16 weeks | 12-16 weeks
  mean change in PHQ9 score with GLP1 receptor agonist over 12-16 weeks (determined at stage 2 by comparing the questionnaire scores from stages 1 and 2). Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
mean change in generalised anxiety disorder assessment (GAD) score with GLP1 receptor agonist over 12-16 weeks | 12-16 weeks
  mean change in GAD score with GLP1 receptor agonist over 12-16 weeks (determined at stage 2 by comparing the questionnaire scores from stages 1 and 2). Score between 0 and 21; scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
mean change in eating disorder examination questionnaire (EDE-Q) score with GLP1 receptor agonist over 12-16 weeks | 12-16 weeks
  mean change in EDE-Q score with GLP1 receptor agonist over 12-16 weeks (determined at stage 2 by comparing the questionnaire scores from stages 1 and 2). Score between 0 and 168, higher scores on the global scale and subscales denote more problematic eating behaviours and attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Khalida Ismail, Principal Investigator — King's College London
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No